CLINICAL TRIAL: NCT04769271
Title: Intra-pocket Application of Tea Tree Oil Gel in the Treatment of Stage-2 Periodontitis (A Clinical and Biochemical Study)
Brief Title: Intra-pocket Application of Tea Tree Oil Gel in the Treatment of Stage-2 Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Maha Talaab, Associate Professor, Oral Medicine, Periodontology, Oral Diagnosis and Oral Radiology department, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tea tree oil & periodontitis
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing; Tea Tree Oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scaling and Root Planing (SRP) (Active Comparator)
  Interventions: Procedure: Scaling and Root Planing
- Scaling and Root Planing with tea tree oil (Experimental)
  Interventions: Drug: Scaling and Root Planing with tea tree oil

INTERVENTIONS:
Procedure: Scaling and Root Planing — Supra- and sub-gingival calculus and debris were removed
  Arms: Scaling and Root Planing (SRP)
Drug: Scaling and Root Planing with tea tree oil — Supra- and sub-gingival calculus and debris were removed and 5% tea tree oil was applied
  Arms: Scaling and Root Planing with tea tree oil

SUMMARY:
This study aimed to assess clinically and biochemically the effect of intrapocket application of tea tree oil (TTO) gel adjunctive to SRP in the management of stage 2(moderate) periodontitis and to correlate the biochemical levels with clinical response.

DETAILED DESCRIPTION:
A randomized, controlled clinical trial included thirty patients with stage 2 periodontitis. They were equally divided into two groups: Group 1 (control group) treated with scaling and root planning (SRP) alone and Group 2 (test group) managed by SRP and locally delivered 5% tea tree oil (TTO) gel.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage 2,grade B periodontitis according to the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions.
* Patients with CAL 3-4 mm , BOP and radiographic horizontal bone loss related to the coronal third of the root (15%-33%).
* Patients with no teeth loss due to periodontitis.
* Patients with radiographic bone loss/age % of 0.25-1 %.
* Patients who could maintain an O'Leary plaque index ≤10 proceeded into the study.

Exclusion Criteria:

* Patients with CAL caused by non periodontal causes.
* Patients with grade C periodontitis.
* Patients having any systemic disease that may affect the treatment outcomes
* Smokers.
* Pregnant females.
* Patients receiving contraindicated medications, chemotherapy, or radiotherapy in the previous year.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Probing depth | up to 6 months
  Probing depth was recorded at tested sites with graduated William's probe graduated in 1 mm increment. Readings were rounded to the nearest mm.
Clinical attachment loss | up to 6 months
  Clinical attachment loss was recorded at tested sites with graduated William's probe graduated in 1 mm increment. Readings were rounded to the nearest mm.
Bleeding on probing | up to 6 months
  Bleeding on probing was assessed at tested sites with graduated William's probe graduated in 1 mm increment, within 15 seconds after probing, using a dichotomous scoring system (+ and -) for presence or absence, respectively.
Biochemical assessment of inlammation | up to 6 months
  This involved determination of the gingival crevicular fluid (GCF) levels of matrix metalloproteinase 8 (MPP-8). A GCF sample was taken from the area showing the deepest pocket depth around the treated area.The samples were diluted in phosphate buffer saline (PBS) up to 1 mL. After waiting for 15 min, the paper points were removed, and 500 μL were centrifuged at 400 g for 4 min, then frozen at -20°C pending MMP-8 analysis using Human Matrix metalloproteinase 8/Neutrophil collagenase (MMP-8) ELISA Kit according to the manufacturer instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Maha R. Taalab, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Dania M. Abdel Aziz, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Sabah A Mahmoud, PhD, Study Director — Medical Biochemistry and Molecular Biology department. Faculty of Dentistry, Alexandria University, Alexandria, Egypt.; Riham M El Moslemany, PhD, Study Director — Pharmaceutics department. Faculty of Pharmacy, Alexandria University; Alexandria, Egypt.
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] Taalab MR, Mahmoud SA, Moslemany RME, Abdelaziz DM. Intrapocket application of tea tree oil gel in the treatment of stage 2 periodontitis. BMC Oral Health. 2021 May 5;21(1):239. doi: 10.1186/s12903-021-01588-y. PMID 33952216